CLINICAL TRIAL: NCT05046938
Title: The Effect of Online Group Motivational Interviewing on Eating Behaviour, Healthy Lifestyle Behaviours and Quality of Life in Nursing Students With Food Addiction: Randomized Controlled Study
Brief Title: Food Addiction and Motivational Interviewing in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Işık (Other)
Responsible Party: Sponsor-Investigator, Merve Işık, research assistant, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Gazi
Record Dates: First submitted 2021-09-01; First posted 2021-09-16 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Food Addiction
Keywords: food addiction; motivational interviewing; healthy life style behaviors; quality of life
MeSH Terms: conditions — Food Addiction | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental design
Who Masked: Investigator
Masking Description: Among the students who meet the food addiction criteria, the students who meet the inclusion criteria and agree to participate in the research will be randomly assigned to the intervention and control groups (n1=29; n2=29). After these students are stratified according to the change (pre-contemplation and contemplation stage) phase, a simple random assignment process within the strata will be done by an independent researcher to avoid selection bias. Random assignment will be done through a simple random numbers table. The independent researcher who does not know which group is the intervention group and which group is the control group will collect the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): It was planned to apply 5 sessions of MI to the intervention group, and to follow-up 2 months after the interviews were completed.
  Interventions: Behavioral: Motivational İnterviewing
- control group (No Intervention): No application will be made to the students in the control group, and at the end of the study, a seminar on food addiction and quality of life will be given to the students.

INTERVENTIONS:
Behavioral: Motivational İnterviewing — Students with food addiction will be provided with motivational interviews about food addiction in 5 sessions, each of which varies between 6-8 groups.
  Arms: intervention group

SUMMARY:
The aim of this study is to determine the effect of online group motivational interviewing (MI) on eating behavior, healthy lifestyle behaviors and quality of life in nursing participants with food addiction at three state universities in Ankara. The population of the research will be those who meet the diagnostic criteria for food addiction according to the Yale Food Addiction Scale. The research sample size was calculated with the G* Power package program. As a result of the power analysis, a total of 52 participants, 26 for the intervention group and 26 for the control group, were found sufficient for the sample with 90% power, 5% margin of error and 0.2065 effect size. Considering that the number of participants would decrease during the research process, the number of samples was increased by 10% to a total of 58 university participants, 29 of which were interventions and 29 were controls. Among the participants who meet the food addiction criteria, the participants who meet the inclusion criteria and agree to participate in the research will be randomly assigned to the intervention and control groups (n1=29; n2=29). After these participants are stratified according to the change (pre-contemplation and contemplation stage) phase, a simple random assignment process within the strata will be done by an independent researcher to avoid selection bias. Random assignment will be done through a simple random numbers table. The independent researcher who does not know which group is the intervention group and which group is the control group will collect the data. Data collection tools will be applied to the participants in the intervention and control groups in the pre-MI session, the post-MI session, and 2 months later in the follow-up session. It was planned to apply 5 sessions of MI to the intervention group, and to follow-up 2 months after the interviews were completed. No application will be made to the participants in the control group, and at the end of the study, a seminar on food addiction and quality of life will be given to the participants.

DETAILED DESCRIPTION:
The research will be conducted as a randomized controlled experimental design to determine the effect of online group motivational interviewing on eating behavior, healthy lifestyle behaviors and quality of life in nursing participants with food addiction.

Research hypotheses:

H0-1: Motivational interview has no effect on the level of healthy lifestyle behaviors of nursing participants.

H1-1: Motivational interview has an effect on the level of healthy lifestyle behaviors of nursing participants.

H0-2: Motivational interview has no effect on the quality of life of nursing students.

H1-2: Motivational interview has an effect on the quality of life of nursing students.

H0-3: Motivational interview has no effect on the eating behavior of nursing students.

H1-3: Motivational interview has an effect on the eating behavior of nursing students.

Place and time of research:

The research will be conducted online on first, second, third and fourth year participants at Gazi University Faculty of Health Sciences Nursing Department, Ankara University Faculty of Nursing and Hacettepe University Faculty of Nursing in the fall semester of the 2021-2022 academic year.

The universe and sample of the research:

Phase One of the Study: The first phase of the study will be carried out between September 2021 and October 2021, after obtaining the ethics committee and institutional permission. There are 635 nurse participants in Ankara University Nursing Faculty, 1022 participants in Hacettepe University Nursing Faculty and 992 nursing participants in Gazi University Faculty of Health Sciences Nursing Department. In order to determine the participants who will be invited to the motivational interview, the "Personal Information Form" and the "Yale Food Addiction Scale" (YFAS) were used as data collection tools for the participants of Ankara University Faculty of Nursing, Hacettepe University Faculty of Nursing and Gazi University Faculty of Health Sciences Nursing Department, to their e-mail addresses and university website. The web-based form will be sent. Participants will first be expected to read the information on the "Participant Informed Consent Form" in the first section and mark the "I Agree" option. After this required field is filled, the data collection tools will be opened for participants to answer the questions. Among the participants who fill in the forms and return to the researcher, those who meet the diagnostic criteria of food addiction according to the YFAS will form the universe of the research. Among the participants who make up the universe, the participants who meet the inclusion criteria of the research will form the sample of the research.

Second Stage of the Research: The sample size of the research was calculated with the calculation (G* Power) package program. In particular, a study that was similar in terms of research design and scale used was examined. The sample calculation for the intervention and control groups planned to be included in the study was based on a study similar to our study. As a result of the power analysis, a total of 52 participants, 26 for the intervention group and 26 for the control group, were found sufficient for the sample with 90% power, 5% margin of error and 0.2065 effect size. Considering that the number of participants would decrease during the research process, the number of samples was increased by 10% and it was increased to a total of 58 university participants, 29 of which were interventions and 29 were controls. Among the participants who meet the food addiction criteria, the participants who meet the inclusion criteria and agree to participate in the research will be randomly assigned to the intervention and control groups (n1=29; n2=29). "The form for determining the stages of change in participants with food addiction" will be applied to the determined participants. After these participants are stratified according to the change (pre-contemplation and contemplation stage) phase, a simple random assignment process within the strata will be done by an independent researcher to avoid selection bias. Random assignment will be done through a simple random numbers table. The independent researcher who does not know which group is the intervention group and which group is the control group will collect the data.

Variables of the Study Independent variables: Motivational interviewing Dependent variables: Quality of life, healthy lifestyle behaviors and eating behavior scales Control (Mixer) Variable: Motivational interview change phase The data of the study will be collected with 'Participant information form', 'Yale Food Addiction Scale', Healthy Lifestyle Behaviors Scale-II and SF-36 Quality of Life Scale.

1. Participant Information Form: Participant information form prepared by the researcher; It consists of a total of 13 questions including socio-demographic characteristics (age, gender, cohabitation, employment status, etc.) and food addiction (height, weight, counseling status) of university participants.
2. Yale Food Addiction Scale (YFAS): The scale, which was developed by Gearhardt et al. in 2009 and adapted into Turkish by Bayraktar et al. in 2012, consists of 27 questions. In the reliability analysis performed for the Food Addiction Scale, the Cronbach's Alpha value of the scale was found to be 0.93. The scale is a scale used to measure addictive-like eating behaviors towards certain types of food (high-fat and high-sugar) in the past 12 months. The scale was created by adapting the substance addiction criteria in DSM-IV to food addiction in order to determine the dependence on specific foods. The first 16 questions of the scale, from 1 to 5, are 'never', 'once a month', 'twice a month', 'twice a week' and 'more than four times a week' and are in a 5-point Likert type. Questions 17-24 will be answered as yes or no. The 25th question includes five items asked about eating habits in the last year. Question 26 includes the preferred nutrient for the nutrition filled by the participant. The 27th question is about whether the person has any other food preferences. The scale is calculated with 7 sub-measures evaluated in the diagnosis of substance addiction. In addition, the scale has an 8th clinical significance score. For the diagnosis of food addiction, at least 3 of the 7 diagnostic criteria must be met and clinical significance must be present. In dystomic scoring, clinical significance, one (1) point of the 15th or 16th item and a symptom score (≥3) are evaluated.
3. Healthy Lifestyle Behaviors Scale-II (HLBS-II): The scale was developed in 1987 as a result of the studies of Walker, Sechrist, and Pender. In 1996, this scale was developed and renamed as the Healthy Lifestyle Behaviors Scale II. The validity and reliability of HLBS- II was established by Bahar et al. in 2008. The cronbach's alpha value of the scale is 0.92 for the total scale, and the reliability coefficients of its sub-dimensions range from 0.64 to 0.80. HLBS II consists of 52 items and six sub-dimensions. Rating is done in the form of a four-point likert. Scale; never (1), sometimes (2), often (3), regularly (4). The lowest score that can be obtained from the scale is 52, and the highest score is 208. Sub-dimensions of the scale; health responsibility, physical activity, nutrition, mental development, interpersonal relationships and stress management.
4. SF-36 Quality of Life Scale: SF-36 was developed by Ware in 1987 for use in the evaluation of clinical practice and health policy in research, and in general population reviews. The scale was translated into Turkish and validity and reliability studies were conducted. The SF-36 was created to provide the minimum psychometric standards required for group comparisons. The items of SF 36 also represent behavioral functions, dysfunctions, and both pleasant and unpleasant personal evaluations such as anxiety and happiness. Each item in the scale is used to score only one subscale. SF 36 is a multi-item measurement tool that evaluates 3 main health areas and 8 health concepts. Among these, physical functionality (10 questions), physical role limitations (4 questions), emotional role limitations (3 questions), social functionality (2 questions) are in functional status. Pain (2 questions), mental health (5 questions), and energy/vitality (4 questions) are included in the field of well-being. General health perception (5 questions) is included in the general assessment of health. There is also an item on the scale that evaluates changes in health during the past year. Except for the fourth and fifth items, the evaluation criterion is likert type, and the fourth and fifth items are answered as yes/no. Subscales evaluate health between 0 and 100, and '0' indicates poor health, while '100' indicates good health.

Application First of all, participants will be expected to answer the "Participant Information Form" and "Yale Food Addiction Scale (YFAS)" respectively. Among the participants who fill in the forms completely and return to the researcher, the participants who meet at least 3 diagnostic criteria according to YFAS and have clinical significance will form the universe of the research. Among the participants who make up the universe, the participants who meet the inclusion criteria of the research will form the sample of the research. The participants who accept to participate in the research will be given the "Identification of Change Stages in participants with Food Addiction Form". According to the change stages, one of the similar groups will be randomly assigned as the intervention group and the other as the control group.

In the second stage of the study, after determining the participants who meet the diagnostic criteria and have clinical significance according to the YFAS, they will be stratified according to the stages of change (pre-contemplation and contemplation) and assigned to the intervention and control groups by an independent researcher with a simple random assignment. A total of 58 participants who want to continue the research will be determined in the intervention and control groups. Data collection tools for the participants in the intervention group who participated in the research between November 2021 and March 2022 before MI session, Week 5 (final session) and 2 months later in the follow-up session. It was planned to apply 5 sessions of motivational interviewing to the intervention group, and to conduct a follow-up interview 2 months after the interviews were completed. The group counseling process will be completed in 5 sessions in total. Group sessions will be held for 60-75 minutes and once a week. Assignment of participants to the groups will be made in line with the limits of the minimum 6 and maximum 8 participants. The day and time of the groups will be determined with the researcher before the first session, outside the class hours of the participants, and the sessions will continue on the same day and time every week. Sessions will be held online. One day before each session, participants will be called by phone and reminded about the time of the session. Data collection tools will be applied to the participants in the control group simultaneously with the first group session, 3 times in the first session, in the 5th week and 2 months later. No application will be made to the participants in the control group, and a webinar will be given to the participants at the end of the study on food addiction and quality of life. An online motivational interview will be held with the participants who make the request. Motivational Interview Plan was created by the researcher and will be submitted to expert opinion. The pre-application researcher participated in the Motivational Interview (MI) training program and received a certificate.

ELIGIBILITY:
Inclusion Criteria:

* Meeting at least 3 diagnostic criteria according to the Yale Food Addiction Scale (YFAS) and having clinical significance
* Not having a written or verbal communication problem
* Volunteer to participate in research
* Among the motivational interview change stages, those who do not intend to change their eating behavior and those who intend to do so

Exclusion Criteria:

* Having a neurological or psychiatric illness that interferes with reading and understanding data collection tools
* Have previously received treatment/psychotherapy for food addiction/eating disorder
* Receiving ongoing treatment/psychotherapy/psychological counseling regarding food addiction/eating disorder
* Having trouble speaking/understanding Turkish
* Being at the stage of preparation, action and maintenance in making changes in nutritional behavior, which is one of the motivational interview change stages

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Evolution of eating behaviour | 5 weeks after randomization
  Yale Food Addiction Scale (Measured by the Yale Food Addiction Scale Minimum score = 0 symptoms, Maximum score = 11 symptoms. Greater symptoms mean worse outcome.

SECONDARY OUTCOMES:
Evolution of health lifestyle behaviour | From baseline, up to 3 months
  Health Lifestyle Behaviour Scale II (Minimum score = 52 score, Maximum score: 208 score.Greater scores mean better outcome.
Evolution of SF-36 quality of life | From baseline, up to 3 months
  SF-36 Quality of Life Scale (Subscales evaluate health between 0 and 100, and '0' indicates poor health, while '100' indicates good health.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Işık, Principal Investigator — Gazi University Faculty of Health Sciences Department of Nursing; Satı Demir, Principal Investigator — Gazi University Faculty of Health Sciences Department of Nursing
Locations (1):
- Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gearhardt AN, Corbin WR, Brownell KD. Preliminary validation of the Yale Food Addiction Scale. Appetite. 2009 Apr;52(2):430-6. doi: 10.1016/j.appet.2008.12.003. Epub 2008 Dec 11. PMID 19121351
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Walker SN, Sechrist KR, Pender NJ. The Health-Promoting Lifestyle Profile: development and psychometric characteristics. Nurs Res. 1987 Mar-Apr;36(2):76-81. PMID 3644262
- [Background] Mokhtari MR, Alavi M, Pahlavanzadeh S, Weimand BM, Visentin D, Cleary M. Comparison of the effectiveness of a 12 step substance use recovery program on quality of life. Nurs Health Sci. 2020 Jun;22(2):390-397. doi: 10.1111/nhs.12668. Epub 2019 Dec 11. PMID 31828941